CLINICAL TRIAL: NCT06161064
Title: Voice and Swallow Outcomes After Office-based Injection Laryngoplasty in Patients With Glottal Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Bakhiet Mahmoud, sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sohagu
Record Dates: First submitted 2023-11-21; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Voice and Swallow Outcomes After Injection Laryngoplasty in Patients With Glottal Insufficiency
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- office-based injection laryngoplasty (Other): office-based injection laryngoplasty by using hyaluronic acid
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Drug: Hyaluronic acid — hyaluronic acid is temporary material using for augmentation of vocal folds in patients with glottal insufficiency

SUMMARY:
The purpose of this study is to evaluate voice quality and swallow outcomes of office-based injection laryngoplasty using hyaluronic acid in patients with Glottal insufficiency and assess all cases after 1, 3 and 6 months.

DETAILED DESCRIPTION:
Glottic insufficiency (incompetence) is characterized by incomplete closure of the vocal folds when phonating, which causes inappropriate leakage of air through the glottis on attempting to phonate and there is an increased risk of aspiration. A wide range of laryngeal symptoms including dysphonia with or without dysphagia may result .There are varieties of causes of glottic insufficiency (GI); among the most common causes of symptomatic GI are vocal fold paralysis (complete immobility of the vocal fold), vocal fold paresis (weakness or partial immobility of the vocal fold) and presbylaryngis. Other causes of GI are sulcus vocalis, scarring or deformation of the vocal folds .Therefore, different therapy options were proposed for patients with GI based on the size of the glottic gap. Voice therapy is most suitable for patients with minimal glottic gap, regardless the reason.Injection augmentation is reserved for those with small or medium-sized glottic gap .Office-based vocal fold injection was used worldwide in early & late Cases of GI. Office-based vocal fold injection in acute cases such as iatrogenic injury of recurrent laryngeal nerve during surgery has many advantages, these include immediate symptomatic relief, the ability to titrate degree of medialization for optimized outcomes, and monitoring of the airway.Moreover, injection in early cases prevent compensatory mechanisms as ventricular hypertrophy. Recent studies suggest that injection laryngoplasty in early cases reduce the need for permanent laryngeal framework surgery.The ideal material to be used for injection should be biocompatible and inert to decrease the risk of local tissue reaction or fibrosis. Also, the material should be easy to use and have a low cost. Furthermore, it should be durable and resistant to resorption or migration, while it maintains the normal viscoelasticity of the vocal cord after injection.

So, there are 2 types of injection materials: temporary &permanent materials. Long-lasting injection materials(permanent) include autologous fat,calcium hydroxylapatite(CaHA) and taflon. Temporary injection materials include bovine gelatin, collagen-based products, carboxymethylcellulose and hyaluronic acid gel (HA). HA is among the most commonly used substances for injection laryngoplasty.

Actually, office-based vocal fold injection has different techniques such as percutaneous (trans-cricothyroid membrane, trans-thyroid cartilage, and trans-thyrohyoid membrane), per-oral, and trans-nasal endoscopic approaches. Typically, the three approaches are performed with a flexible laryngoscope in place, visualizing the larynx for visualization and to monitor injection effects.

ELIGIBILITY:
Inclusion Criteria:

1. The complaint of all patients is dysphonia with or without aspiration
2. Patients with small or large glottic gap
3. Patients at least 1-2 months after the onset of GI

Exclusion Criteria:

Patients who are 1- >18 years old 2-Irritable 3-Exaggerated gag reflexes 4-Cardiac problems 5-Active laryngeal carcinoma 6-Patients on chemo or radiotherapy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
voice evaluation using voice handicap index in patients with glottal insufficiency before and after injection laryngoplasty | 1, 3 and 6 months
  voice handicap index is a multiple questions about voice disorders patients answered before and after injection laryngoplasty

SECONDARY OUTCOMES:
voice evaluation using acoustics in patients with glottal insufficiency before and after injection laryngoplasty | 1, 3 and 6 months
  The vocal samples are obtained from the participants by holding a Microphone 10 cm in front of their mouth and producing sustained phonation. Each participant is asked to sustain the vowels /a/ /i/ /u/ followed by connected speech (counting from 1-5) using habitual and constant vocal pitch, loudness, and quality for at least 5 seconds with elimination of the irregularities in the beginning and end of utterance. The room for sampling is situated away from noise. Acoustic parameters as: Fundamental frequency, Jitter, Shimmer and noise to harmonic ratio

CONTACTS AND LOCATIONS:
Overall Officials: ayaa bakhet, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: Yes
voice and swallow outcomes after office-based injection laryngoplasty in patients with glottal insufficiency
Supporting Information: SAP
Time Frame: december,2024